CLINICAL TRIAL: NCT03617523
Title: Safety and Immunogenicity of Fluzone® Quadrivalent, Flublok® Quadrivalent, and Fluzone® High-Dose, Influenza Vaccines, 2018-2019 Formulations
Acronym: GRC90
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC90; U1111-1211-4864 (Other: UTN)
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: The study was partially randomized. Participants were assigned a vaccine group based on age. Participants in Groups 1, 2, and 5 were not randomly assigned, while participants in Groups 3 and 4 were randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Fluzone Quadrivalent vaccine Group 1: 6 to <36 months (Experimental): Participants (aged 6 to <36 months) received a 0.25-milliliter (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2018-2019 formulation
- Fluzone Quadrivalent vaccine Group 2: 3 to <9 years (Experimental): Participants (aged 3 to <9 years) received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2018-2019 formulation
- Fluzone Quadrivalent vaccine Group 3: 18 to <65 years (Experimental): Participants (aged 18 to <65 years) received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2018-2019 formulation
- Flublok Quadrivalent vaccine Group 4: 18 to <65 years (Experimental): Participants (aged 18 to <65 years) received a 0.5-mL dose of Flublok Quadrivalent vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Flublok Quadrivalent vaccine, 2018-2019 formulation
- Fluzone High-Dose vaccine Group 5: >=65 years (Experimental): Participants (aged >=65 years) received a 0.5-mL dose of Fluzone High-Dose vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone High-Dose vaccine, 2018-2019 formulation

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, 2018-2019 formulation — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Fluzone Quadrivalent vaccine Group 1: 6 to <36 months; Fluzone Quadrivalent vaccine Group 2: 3 to <9 years; Fluzone Quadrivalent vaccine Group 3: 18 to <65 years
Biological: Flublok Quadrivalent vaccine, 2018-2019 formulation — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Flublok Quadrivalent vaccine Group 4: 18 to <65 years
Biological: Fluzone High-Dose vaccine, 2018-2019 formulation — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Fluzone High-Dose vaccine Group 5: >=65 years

SUMMARY:
The primary objectives of this study were:

* To describe the immunogenicity of the 2018-2019 formulation of Fluzone® Quadrivalent vaccine in children 6 to less than (<) 36 months of age and 3 to <9 years of age, and in adults 18 to <65 years of age; the immunogenicity of the 2018-2019 formulation of Flublok® Quadrivalent vaccine in adults 18 to <65 years of age; and the immunogenicity of the 2018-2019 formulation of Fluzone High-Dose vaccine in adults greater than or equal to (>=) 65 years of age.
* To describe the safety of the 2018-2019 formulation of Fluzone Quadrivalent vaccine in children 6 to <36 months of age and 3 to <9 years of age, and in adults 18 to <65 years of age; the safety of the 2018-2019 formulation of Flublok Quadrivalent vaccine in adults 18 to <65 years of age; and the safety of the 2018-2019 formulation of Fluzone High-Dose vaccine in adults >=65 years of age.

DETAILED DESCRIPTION:
Study duration per participant was approximately 21 days for adult participants or 28 days for child participants who received one dose of vaccine, and 56 days for participants who received two doses of vaccine.

ELIGIBILITY:
Inclusion criteria :

* Aged 6 months to <9 years or >=18 years on the day of first study vaccination (study product administration).
* For participants 6 to <12 months of age, born at full term of pregnancy (>=37 weeks) and with a birth weight >=2.5 kilograms (kg) (5.5 pounds [lbs.]).
* Informed consent form (ICF) had been signed and dated by participants >=18 years of age.
* Assent form had been signed and dated by participants 7 to <9 years of age, and ICF had been signed and dated by parent(s) or guardian(s) for participants 6 months to <9 years of age.
* Participants and parent/guardian (of participants 6 months to <9 years of age) were able to attend all scheduled visits and to comply with all study procedures.

Exclusion criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 30 days preceding the first study vaccination, or planned receipt of any vaccine before Visit 2 for participants who received 1 dose of influenza vaccine or Visit 3 for participants who received 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2018-2019 influenza season) with either study vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the 3 months preceding planned inclusion.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the 6 months preceding planned inclusion; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life- threatening reaction to study vaccine or to a vaccine containing any of the same substances.
* Thrombocytopenia, which might be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature >=100.4 degree Fahrenheit [38.0 degree Celsius]). A prospective participant was not included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study (participants >=18 years of age) or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study (all participants).
* History of serious adverse reaction to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- United States (3):
  - Investigational Site Number 8400003, Bardstown, Kentucky
  - Investigational Site Number 8400001, Metairie, Louisiana
  - Investigational Site Number 8400002, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 10 September 2018 to 22 October 2018 at 3 centers in the United States.
Pre-assignment Details: A total of 240 participants were enrolled in the study.
Groups:
- Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months: Participants (aged 6 to less than [<] 36 months) received a 0.25-milliliter (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Fluzone High-Dose Vaccine Group 5: >=65 Years: Participants (aged greater than or equal to [>=] 65 years) received a 0.5-mL dose of Fluzone High-Dose vaccine, intramuscularly, at Day 0.
Period: Overall Study
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
Started | 30 | 30 | 61 | 59 | 60
Completed | 30 | 30 | 61 | 59 | 60
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety analysis set which included participants who received at least 1 dose of study vaccine.
Groups:
- Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months: Participants (aged 6 to <36 months) received a 0.25-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Total: Total of all reporting groups
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years | Total
Number analyzed (Participants) | 30 | 30 | 61 | 59 | 60 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.7 (0.44) | 5.9 (1.76) | 46.7 (13.48) | 46.2 (13.44) | 73.6 (6.42) | 42.6 (26.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 45 | 42 | 40 | 152
  Male | 17 | 18 | 16 | 17 | 20 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 20 | 12 | 4 | 54
  White | 18 | 19 | 41 | 46 | 56 | 180
  More than one race | 3 | 2 | 0 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Group 1: Aged 6 to <36 Months) Reporting Solicited Injection Site Reactions and Systemic Reactions
Description: A solicited reaction was an adverse event (AE) that was pre-listed in the electronic case report form (eCRF) and considered to be related to vaccination. Solicited injection (Inj.) site reactions: tenderness, erythema and swelling. Solicited systemic reactions: fever, vomiting, crying abnormal, drowsiness, appetite lost and irritability.
Time Frame: Within 7 days post any vaccination
Population: Analysis was performed on safety analysis set. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months
Number analyzed (Participants) | 29
Participants
  Injection site tenderness | 15
  Injection site erythema | 3
  Injection site swelling | 4
  Fever | 2
  Vomiting | 3
  Crying abnormal | 4
  Drowsiness | 9
  Appetite lost | 10
  Irritability | 12

2. Primary Outcome: Number of Participants (Groups 2, 3, 4 and 5: Children Aged 3 to <9 Years and Adults 18 to >=65 Years) Reporting Solicited Injection Site Reactions or Systemic Reactions
Description: A solicited reaction was an AE that was pre-listed in the eCRF and considered to be related to vaccination. Solicited injection site reactions: pain, erythema and swelling. Solicited systemic reactions: fever, headache, malaise, and myalgia.
Time Frame: Within 7 days post any vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
Number analyzed (Participants) | 30 | 61 | 59 | 60
Participants
  Injection site pain | 9 | 27 | 22 | 24
  Injection site erythema | 5 | 1 | 0 | 5
  Injection site swelling | 6 | 2 | 0 | 3
  Fever | 1 | 0 | 0 | 0
  Headache | 5 | 12 | 13 | 11
  Malaise | 6 | 11 | 6 | 9
  Myalgia | 6 | 14 | 11 | 15

3. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies in Children 6 Months to <9 Years of Age (Groups 1 and 2) Receiving Fluzone Quadrivalent Vaccine
Description: GMT of anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage.
Time Frame: 28 days post-final vaccination
Population: Analysis was performed on per-protocol analysis set which included participants who received at least 1 dose of the study vaccine and had a valid post-vaccination blood sample result for at least 1 strain without any protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years
Number analyzed (Participants) | 26 | 29
titers (1/dilution)
  A/H1N1 | 229 [108 to 487] | 1008 [605 to 1680]
  A/H3N2 | 239 [94.0 to 606] | 1109 [671 to 1833]
  B Victoria | 160 [79.3 to 323] | 688 [390 to 1211]
  B Yamagata | 295 [167 to 524] | 1343 [811 to 2223]

4. Primary Outcome: Geometric Mean Titers of Antibodies in Adults (Groups 3, 4 and 5) Receiving Either Fluzone Quadrivalent Vaccine, Flublok Quadrivalent Vaccine, or Fluzone High-Dose Vaccine
Description: GMTs of anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage in Groups 3 and 4, and using HAI assay for 3 strains: A/H1N1, A/H3N2 and B Victoria lineage in Group 5.
Time Frame: Day 21 (post-vaccination)
Population: Analysis was performed on per-protocol analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilutions)
Arm/Group | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
Number analyzed (Participants) | 61 | 58 | 60
titers (1/dilutions)
  A/H1N1 | 525 [386 to 712] | 708 [498 to 1007] | 266 [195 to 363]
  A/H3N2 | 379 [276 to 523] | 644 [456 to 909] | 359 [255 to 507]
  B Victoria | 588 [447 to 773] | 525 [388 to 711] | 453 [337 to 608]
  B Yamagata | 759 [571 to 1009] | 1102 [829 to 1465] | NA [NA to NA] — Data not reported since the immune response to the B Yamagata lineage strain was not assessed in Group 5 participants.

5. Primary Outcome: Geometric Mean Titer Ratios (GMTRs) of Antibodies in Children 6 Months to <9 Years of Age (Groups 1 and 2) Receiving Fluzone Quadrivalent Vaccine
Description: GMT of anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage. GMTRs were calculated as the ratio of GMTs post-final vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination), 28 days post-final vaccination
Population: Analysis was performed on per-protocol analysis set. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years
Number analyzed (Participants) | 25 | 28
ratio
  A/H1N1(post-final vaccination/pre-vaccination) | 9.06 [5.38 to 15.3] | 4.47 [2.39 to 8.35]
  A/H3N2(post-final vaccination/pre-vaccination) | 3.94 [1.92 to 8.12] | 6.40 [3.95 to 10.4]
  B Victoria(post-final vaccination/pre-vaccination) | 8.11 [4.84 to 13.6] | 13.3 [8.61 to 20.5]
  B Yamagata(post-final vaccination/pre-vaccination) | 11.8 [7.24 to 19.2] | 8.41 [4.98 to 14.2]

6. Primary Outcome: Geometric Mean Titer Ratios of Antibodies in Adults (Groups 3, 4 and 5) Receiving Either Fluzone Quadrivalent Vaccine, Flublok Quadrivalent Vaccine, or Fluzone High-Dose Vaccine
Description: GMTs of anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage in Groups 3 and 4, and using HAI assay for 3 strains: A/H1N1, A/H3N2 and B Victoria lineage in Group 5. GMTRs were calculated as the ratio of GMTs post vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination), Day 21 (post-vaccination)
Population: Analysis was performed on per-protocol analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
Number analyzed (Participants) | 61 | 58 | 60
ratio
  A/H1N1 (post-vaccination/pre-vaccination) | 2.93 [2.02 to 4.23] | 6.34 [4.17 to 9.63] | 3.07 [2.34 to 4.02]
  A/H3N2 (post-vaccination/pre-vaccination) | 3.55 [2.60 to 4.85] | 8.19 [5.56 to 12.1] | 3.69 [2.68 to 5.08]
  B Victoria (post-vaccination/pre-vaccination) | 3.39 [2.43 to 4.73] | 4.40 [3.13 to 6.19] | 3.65 [2.79 to 4.76]
  B Yamagata (post-vaccination/pre-vaccination) | 2.84 [2.10 to 3.85] | 5.20 [3.76 to 7.21] | NA [NA to NA] — Data not reported since the immune response to the B Yamagata lineage strain was not assessed in Group 5 participants.

7. Primary Outcome: Percentage of Participants With Seroprotection to Influenza Vaccine Antigens After Vaccination With Fluzone Quadrivalent Vaccine: Groups 1 and 2
Description: Anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage. Seroprotection was defined as antibody titer >=40 (1/ dilution) at pre-vaccination and at post-final vaccination.
Time Frame: 28 days post-final vaccination
Population: Analysis was performed on per-protocol analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years
Number analyzed (Participants) | 26 | 29
percentage of participants
  A/H1N1 | 84.6 [65.1 to 95.6] | 96.6 [82.2 to 99.9]
  A/H3N2 | 80.8 [60.6 to 93.4] | 96.6 [82.2 to 99.9]
  B Victoria | 80.8 [60.6 to 93.4] | 100 [88.1 to 100]
  B Yamagata | 92.3 [74.9 to 99.1] | 96.6 [82.2 to 99.9]

8. Primary Outcome: Percentage of Participants With Seroprotection to Influenza Vaccine Antigens After Vaccination With Either Fluzone Quadrivalent Vaccine, Flublok Quadrivalent Vaccine or Fluzone High Dose Vaccine: Group 3, 4 and 5
Description: Anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage in Groups 3 and 4, and using HAI assay for 3 strains: A/H1N1, A/H3N2 and B Victoria lineage in Group 5. Seroprotection was defined as antibody titer >=40 (1/dilution) at pre-vaccination and at post-final vaccination.
Time Frame: Day 21 (post-vaccination)
Population: Analysis was performed on per-protocol analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
Number analyzed (Participants) | 61 | 58 | 60
percentage of participants
  A/H1N1 | 100 [94.1 to 100] | 100 [93.8 to 100] | 93.3 [83.8 to 98.2]
  A/H3N2 | 98.4 [91.2 to 100] | 100 [93.8 to 100] | 98.3 [91.1 to 100]
  B Victoria | 100 [94.1 to 100] | 98.3 [90.8 to 100] | 98.3 [91.1 to 100]
  B Yamagata | 100 [94.1 to 100] | 100 [93.8 to 100] | NA [NA to NA] — Data not reported since the immune response to the B Yamagata lineage strain was not assessed in Group 5 participants.

9. Primary Outcome: Percentage of Participants With Seroconversion to Influenza Vaccine Antigens After Vaccination With Fluzone Quadrivalent Vaccine: Group 1 and 2
Description: Anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage. Seroconversion was defined as either a pre-vaccination titer <10 (1/dilution) and a post-final vaccination titer >= 40 (1/dilution) or a pre-vaccination titer >= 10 (1/dilution) and >=4-fold increase in post-final vaccination titer.
Time Frame: 28 days post-final vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years
Number analyzed (Participants) | 25 | 28
percentage of participants
  A/H1N1 | 80.0 [59.3 to 93.2] | 42.9 [24.5 to 62.8]
  A/H3N2 | 56.0 [34.9 to 75.6] | 64.3 [44.1 to 81.4]
  B Victoria | 80.0 [59.3 to 93.2] | 92.9 [76.5 to 99.1]
  B Yamagata | 88.0 [68.8 to 97.5] | 78.6 [59.0 to 91.7]

10. Primary Outcome: Percentage of Participants With Seroconversion to Influenza Vaccine Antigens After Vaccination With Either Fluzone Quadrivalent Vaccine, Flublok Quadrivalent Vaccine or Fluzone High Dose Vaccine: Group 3, 4 and 5
Description: Anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage in Group 3 and 4, and using an HAI assay for 3 strains: A/H1N1, A/H3N2, and B Victoria lineage in Group 5. Seroconversion was defined as either a pre-vaccination titer <10 (1/dilution) and a post-vaccination titer >= 40 (1/dilution) or a pre-vaccination titer >= 10 (1/dilution) and >=4-fold increase in post-vaccination titer.
Time Frame: Day 21 (post-vaccination)
Population: Analysis was performed on per-protocol analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Fluzone High-Dose Vaccine Group 5: >=65 Years: Participants (aged >=65 years) received a 0.5-mL dose of Fluzone High-Dose vaccine, intramuscularly, at Day 0.
  .
Arm/Group | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
Number analyzed (Participants) | 61 | 58 | 60
percentage of participants
  A/H1N1 | 32.8 [21.3 to 46.0] | 51.7 [38.2 to 65.0] | 46.7 [33.7 to 60.0]
  A/H3N2 | 44.3 [31.5 to 57.6] | 70.7 [57.3 to 81.9] | 50.0 [36.8 to 63.2]
  B Victoria | 32.8 [21.3 to 46.0] | 46.6 [33.3 to 60.1] | 46.7 [33.7 to 60.0]
  B Yamagata | 27.9 [17.1 to 40.8] | 55.2 [41.5 to 68.3] | NA [NA to NA] — Data not reported since the immune response to the B Yamagata lineage strain was not assessed in Group 5 participants.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 0 (post-vaccination) up to study end ( i.e., up to Day 21 for adult participants or Day 28 for child participants who received 1 dose; up to Day 56 for participants who received 2 doses).
Description: Solicited reaction (SR) is an AE prelisted in eCRF and considered related to vaccination. A SR is, therefore, an adverse drug reaction observed and reported under conditions prelisted (solicited) in eCRF. An Unsolicited AE is an observed AE that does not fulfill conditions prelisted in eCRF in terms of symptom and/or time to onset post-vaccination. Non-serious adverse events (non-SAE) included SR (within 7 days after vaccination) and unsolicited non-SAE (within 28 days after final vaccination)
Groups:
- Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months: Participants (aged 6 to <36 months) received a 0.25 mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years: Participants (aged 3 to <9 years) received a 0.5 mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years: Participants (aged 18 to <65 years) received a 0.5 mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0.
- Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years: Participants (aged 18 to <65 years) received a 0.5 mL dose of Flublok Quadrivalent vaccine, intramuscularly, at Day 0.
- Fluzone High-Dose Vaccine Group 5: >=65 Years: Participants (aged >=65 years) received a 0.5 mL dose of Fluzone High-Dose vaccine, intramuscularly, at Day 0.
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years | Fluzone High-Dose Vaccine Group 5: >=65 Years
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/61 | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/61 | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 21/30 | 13/30 | 33/61 | 29/59 | 34/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Quadrivalent Vaccine Group 1: 6 to <36 Months (N=30) | Fluzone Quadrivalent Vaccine Group 2: 3 to <9 Years (N=30) | Fluzone Quadrivalent Vaccine Group 3: 18 to <65 Years (N=61) | Flublok Quadrivalent Vaccine Group 4: 18 to <65 Years (N=59) | Fluzone High-Dose Vaccine Group 5: >=65 Years (N=60)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crying (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 5 (5)
Injection Site Pain (General disorders) | 15 (16) | 9 (9) | 27 (27) | 22 (22) | 24 (24)
Injection Site Swelling (General disorders) | 4 (5) | 6 (6) | 2 (2) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 6 (6) | 11 (11) | 6 (6) | 9 (9)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 15 (15) | 11 (11) | 15 (15)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 12 (12) | 14 (15) | 11 (11)
Somnolence (Nervous system disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 12 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03617523/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03617523/SAP_001.pdf